CLINICAL TRIAL: NCT04251364
Title: Acetazolamide and Statins for the Treatment of Chronic Mountain Sickness in Highlanders: A Randomized Controlled Trial
Brief Title: Treatment of Chronic Mountain Sickness
Acronym: Exp5300
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Expertise sur l'Altitude EXALT (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Expedition5300
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hypoxia, Altitude
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acetazolamide (Experimental): Oral acetazolamide (250 mg/day) intake for 9 months
  Interventions: Drug: Acetazolamide
- Atorvastatin (Experimental): Oral atorvastatin (40 mg/day) intake for 9 months
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Oral placebo pill (daily) intake for 9 months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Acetazolamide — Daily acetazolamide pill intake
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Atorvastatin — Daily atorvastatin pill intake
  Arms: Atorvastatin
Drug: Placebo oral tablet — Daily placebo pill intake
  Arms: Placebo

SUMMARY:
This study aims to assess the effect of two drugs for the treatment of chronic mountain sickness in highlanders.

DETAILED DESCRIPTION:
About 100 million individuals reside at high altitude (>2500m) worldwide, with the largest populations of highlanders being found in South America (Andean), central Asia (Tibetan and Sherpa) and East Africa (Ethiopian). Despite unique adaptations to hypoxia in these populations, chronic mountain sickness (CMS) is a clinical syndrome which is observed in 5-33% of individuals residing permanently at high altitude.Several pharmacological approaches have been proposed in the treatment of EE and CMS. However, few studies show sufficient clinical evidence for safety and efficacy in CMS treatment and most highlanders with CMS remain untreated. The present project aims to better characterize chronic hypoxic responses in highlanders and to evaluate the interest of acetazolamide and statins as potential treatments for chronic mountain sickness.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 55 yrs
* Body mass index <30kg/m²
* Born at >3500 m, living for >3 years at the local high altitude
* No diagnosis of cardiorespiratory, metabolic or neurological diseases
* No drug intake
* No smoker
* Chronic mountain sickness score ≥6

Exclusion Criteria:

* Diagnosis of cardiorespiratory, metabolic and neurological diseases
* Systolic > 130 mmHg and/or diastolic > 85 mmHg blood pressure
* Drug intake
* Smoker
* Chronic mountain sickness score <6

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in hematocrit | Change from before to after 9 months of treatment
  Change in blood hematocrit value in percentage

SECONDARY OUTCOMES:
Chronic mountain sickness score | Change from before to after 9 months of treatment
  Chronic mountain sickness score (between 0 and 24, the higher the score the more severe the sickness) according to the available international scoring system
Macrovascular reactivity | Change from before to after 9 months of treatment
  Post-ischemia brachial artery dilation in %
Microvascular reactivity | Change from before to after 9 months of treatment
  Hyperthermic microvascular dilation in %
Hemoglobin mass | Change from before to after 9 months of treatment
  Total blood hemoglobin mass in mg
Pulmonary arterial pressure | Change from before to after 9 months of treatment
  Systolic and mean pulmonary arterial pressure in mmHg
Blood pressure | Change from before to after 9 months of treatment
  24-hour systolic and diastolic blood pressure
Sleep recording | Change from before to after 9 months of treatment
  Hypopnea-apnea index reported in number of events per hour

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Verges, PhD, Principal Investigator — EXAL
Locations (1):
- Association EXALT, UM Sport Pathologies, Hôpital Sud, Avenue Kimberley, Échirolles, France

IPD SHARING:
Plan to Share IPD: No